CLINICAL TRIAL: NCT06045507
Title: A Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral MK-8527 Once Monthly in Participants at Low-Risk for HIV-1 Infection
Brief Title: Safety and Pharmacokinetic Study of Oral MK-8527 QM in Participants at Low-Risk for HIV-1 Infection (MK-8527-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8527-007
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Results first posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: HIV; HIV Pre-exposure Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MK-8527 Low Dose QM (Experimental): Participants receive oral MK-8527 low dose QM for 6 months, followed by an 8-week blinded safety follow-up period.
  Interventions: Drug: MK-8527
- MK-8527 Medium Dose QM (Experimental): Participants receive oral MK-8527 medium dose QM for 6 months, followed by an 8-week blinded safety follow-up period.
  Interventions: Drug: MK-8527
- MK-8527 High Dose QM (Experimental): Participants receive oral MK-8527 high dose QM for 6 months, followed by an 8-week blinded safety follow-up period.
  Interventions: Drug: MK-8527
- Placebo to MK-8527 (Placebo Comparator): Participants receive oral placebo matched to MK-8527 QM for 6 months, followed by an 8-week blinded safety follow-up period.
  Interventions: Drug: Placebo to MK-8527

INTERVENTIONS:
Drug: MK-8527 — MK-8527 capsule
  Arms: MK-8527 High Dose QM; MK-8527 Low Dose QM; MK-8527 Medium Dose QM
Drug: Placebo to MK-8527 — Placebo capsule matched to MK-8527
  Arms: Placebo to MK-8527

SUMMARY:
This double-blind, placebo-controlled study was designed to assess the safety, tolerability, and pharmacokinetics of oral MK-8527 taken once monthly (QM) in participants at low risk for human immunodeficiency virus Type 1 (HIV-1) infection.

ELIGIBILITY:
Inclusion Criteria:

* Is confirmed HIV-uninfected based on negative HIV-1/HIV-2 test result before randomization
* Has low-risk of HIV infection
* Females: is not pregnant or breastfeeding and is either not a participant of childbearing potential (POCBP) OR is a POCBP and uses an acceptable contraception or is abstinent from penile-vaginal intercourse

Exclusion Criteria:

* Has hypersensitivity or other contraindication to any of the components of the study interventions as determined by the investigator
* Has an active diagnosis of hepatitis due to any cause, including active hepatitis B (HBV) infection (defined as HBsAg-positive) or hepatitis C virus (HCV) infection (defined as detectable HCV ribonucleic acid [RNA])
* Prior use of MK-8527 or islatravir (MK-8591)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (18):
- United States (10):
  - Velocity Clinical Research, North Hollywood ( Site 0054), North Hollywood, California
  - Bridge HIV- San Francisco Department of Public Health ( Site 0042), San Francisco, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0052), Hallandale, Florida
  - Community Medical Care Center ( Site 0056), Immokalee, Florida
  - Velocity Clinical Research Rockville ( Site 0048), Rockville, Maryland
  - Fenway Health ( Site 0043), Boston, Massachusetts
  - Albuquerque Clinical Trials, Inc. ( Site 0044), Albuquerque, New Mexico
  - University of Pittsburgh Medical Center-Division of Infectious Diseases ( Site 0041), Pittsburgh, Pennsylvania
  - Prism Health North Texas, Oak Cliff Health Center ( Site 0045), Dallas, Texas
  - Fred Hutchinson Cancer Center - The Seattle HIV Vaccine Trials Unit ( Site 0057), Seattle, Washington
- Israel (3):
  - Rambam Health Care Campus ( Site 0003), Haifa
  - Hadassah Medical Center ( Site 0002), Jerusalem
  - Sheba Medical Center ( Site 0001), Ramat Gan
- South Africa (5):
  - Josha Research ( Site 0023), Bloemfontein, Free State
  - Wits RHI-Wits RHI Ward 21 Clinical Research site ( Site 0027), Johannesburg, Gauteng
  - Helen Joseph Hospital ( Site 0024), Johannesburg, Gauteng
  - Qhakaza Mbokodo Research Clinic ( Site 0026), Ladysmith, KwaZulu-Natal
  - Desmond Tutu Health Foundation ( Site 0021), Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants who were at low risk of human immunodeficiency virus Type 1 (HIV-1) infection were recruited.
Groups:
- MK-8527 3 mg QM: Participants received oral MK-8527 3 mg once monthly (QM) for 6 months, followed by an 8-week blinded safety follow-up period.
- MK-8527 6 mg QM: Participants received oral MK-8527 6 mg QM for 6 months, followed by an 8-week blinded safety follow-up period.
- MK-8527 12 mg QM: Participants received oral MK-8527 12 mg QM for 6 months, followed by an 8-week blinded safety follow-up period.
- Placebo to MK-8527: Participants received oral placebo matched to MK-8527 QM for 6 months, followed by an 8-week blinded safety follow-up period.
Period: Overall Study
Arm/Group | MK-8527 3 mg QM | MK-8527 6 mg QM | MK-8527 12 mg QM | Placebo to MK-8527
Started | 101 | 102 | 100 | 49
Completed | 92 | 97 | 98 | 46
Not Completed | 9 | 5 | 2 | 3
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 3 | 0 | 0
Not completed — Randomized by mistake (no study treatment given) | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 1 | 0 | 2
Not completed — Miscellaneous | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- MK-8527 3 mg QM: Participants received oral MK-8527 3 mg QM for 6 months, followed by an 8-week blinded safety follow-up period.
- Total: Total of all reporting groups
Arm/Group | MK-8527 3 mg QM | MK-8527 6 mg QM | MK-8527 12 mg QM | Placebo to MK-8527 | Total
Number analyzed (Participants) | 101 | 101 | 99 | 49 | 350
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.4 (10.12) | 30.0 (9.80) | 29.6 (8.84) | 29.8 (8.90) | 30.0 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 58 | 29 | 204
  Male | 43 | 42 | 41 | 20 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 13 | 14 | 11 | 56
  Not Hispanic or Latino | 83 | 86 | 84 | 38 | 291
  Unknown or Not Reported | 0 | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 3 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 44 | 40 | 40 | 21 | 145
  White | 49 | 54 | 51 | 26 | 180
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 5 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥1 Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to ~28 weeks
Population: All randomized participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8527 3 mg QM | MK-8527 6 mg QM | MK-8527 12 mg QM | Placebo to MK-8527
Number analyzed (Participants) | 101 | 101 | 99 | 49
Participants | 62 | 69 | 66 | 31

2. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Dosing to Last Measurable Concentration (AUC0-last) of MK-8527
Description: The plasma AUC0-last of MK-8527 is reported.
Time Frame: Day 1: predose and 0.5, 4, and 24 hours postdose. Week 20: 0.5, 4, and 24 hours postdose
Population: Participants treated with active MK-8527 who complied with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model, are included.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µmol/L
Arm/Group | MK-8527 3 mg QM | MK-8527 6 mg QM | MK-8527 12 mg QM | Placebo to MK-8527
Number analyzed (Participants) | 95 | 96 | 97 | 0
hr*µmol/L
  Day 1 | 0.132 (84.8) | 0.397 (36.1) | 0.861 (34.1) |
  Week 20: number analyzed (Participants) | 78 | 92 | 95 | 0
  Week 20 | 0.129 (81.5) | 0.404 (37.3) | 0.836 (55.0) |

3. Primary Outcome: Number of Participants Discontinuing Study Therapy Due to Adverse Event (AE)
Description: as for outcome 1
Time Frame: Up to ~20 weeks
Population: All randomized participants who received ≥1 dose of study therapy are included.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-8527 3 mg QM | MK-8527 6 mg QM | MK-8527 12 mg QM | Placebo to MK-8527
Number analyzed (Participants) | 101 | 101 | 99 | 49
Participants | 0 | 2 | 1 | 2

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MK-8527
Description: The plasma Cmax of MK-8527 is reported.
Time Frame: Day 1: predose and 0.5, 4, and 24 hours postdose. Week 20: 0.5, 4, and 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µmol/L
Arm/Group | MK-8527 3 mg QM | MK-8527 6 mg QM | MK-8527 12 mg QM | Placebo to MK-8527
Number analyzed (Participants) | 95 | 96 | 97 | 0
µmol/L
  Day 1 | 0.0289 (69.0) | 0.0490 (75.6) | 0.113 (64.5) |
  Week 20: number analyzed (Participants) | 78 | 92 | 95 | 0
  Week 20 | 0.0320 (67.5) | 0.0538 (73.5) | 0.108 (72.5) |

ADVERSE EVENTS:
Time Frame: Up to ~28 weeks
Description: All randomized participants who received ≥1 dose of study therapy are included.
Arm/Group | MK-8527 3 mg QM | MK-8527 6 mg QM | MK-8527 12 mg QM | Placebo to MK-8527
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/101 | 1/99 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/101 | 0/101 | 1/99 | 1/49
Other Adverse Events (participants affected / at risk) | 38/101 | 43/101 | 32/99 | 21/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8527 3 mg QM (N=101) | MK-8527 6 mg QM (N=101) | MK-8527 12 mg QM (N=99) | Placebo to MK-8527 (N=49)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8527 3 mg QM (N=101) | MK-8527 6 mg QM (N=101) | MK-8527 12 mg QM (N=99) | Placebo to MK-8527 (N=49)
Nausea (Gastrointestinal disorders) | 4 (4) | 8 (9) | 3 (3) | 1 (2)
Fatigue (General disorders) | 5 (7) | 8 (11) | 7 (7) | 3 (3)
COVID-19 (Infections and infestations) | 2 (2) | 4 (4) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 16 (19) | 10 (11) | 10 (11) | 6 (8)
Blood creatine phosphokinase increased (Investigations) | 3 (5) | 1 (1) | 3 (3) | 3 (3)
CD4 lymphocytes decreased (Investigations) | 4 (4) | 3 (3) | 5 (6) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 6 (6) | 1 (2)
Headache (Nervous system disorders) | 9 (9) | 7 (7) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (7) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (2):
  • Study Protocol (2024-10-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT06045507/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT06045507/SAP_001.pdf